CLINICAL TRIAL: NCT06092983
Title: A Randomized, Double-Blind, Placebo Controlled, Phase Ib Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple-Dose Escalation HS-10383 in Healthy Adult Subjects
Brief Title: A Multiple-Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetic of HS-10383
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10383-102
Record Dates: First submitted 2023-05-30; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-05

CONDITIONS: Cough
Keywords: RUCC, P2X3
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10383 (Multiple doses) (Experimental): Escalating doses of HS-10383 administered orally once daily for a week in healthy participants.
  Interventions: Drug: HS-10383
- HS-10383 Placebo (Multiple doses) (Placebo Comparator): Escalating doses of HS-10383 Placebo administered orally daily for a week in healthy participants.
  Interventions: Drug: HS-10383 Placebo

INTERVENTIONS:
Drug: HS-10383 — HS-10383 administered as one 50 mg, 150 mg, 300 mg and 450 mg capsule once daily, depending upon randomization.
  Other Names: HS-10383 Tablets
  Arms: HS-10383 (Multiple doses)
Drug: HS-10383 Placebo — HS-10383 Placebo administered as one 50 mg, 150 mg, 300 mg and 450 mg capsule once daily, depending upon randomization.
  Other Names: HS-10383 Placebo Tablets
  Arms: HS-10383 Placebo (Multiple doses)

SUMMARY:
This study will investigate the safety, tolerability and pharmacokinetics of ascending multiple doses of HS-10383 in healthy subjects using a randomized, double blind, placebo controlled, single center study design.

DETAILED DESCRIPTION:
HS-10383 is a selective P2X3 receptor antagonist being developed for the treatment of refractory/unexplained chronic cough. This Phase 1b study will investigate the safety, tolerability and pharmacokinetics of ascending multiple doses of HS-10383 administered orally to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants aged from 18 to 45 years
2. Subjects need to fully understand the research content and process, as well as possible adverse reactions, and voluntarily sign the informed consent;
3. Male weight ≥ 50kg, female weight ≥ 45kg, body mass index {BMI, BMI=weight/height 2 (kg/m2)} is controlled within the range of 18~26 (including the critical value);

Exclusion Criteria:

1. The following medical histories, such as neuropsychiatric system, cardiovascular system, urinary system, digestive system, respiratory system, skeletal muscle system, metabolic endocrine system, skin disease, blood system, immune system and tumor, etc., were screened. evaluated as unsuitable to participate in this study;
2. Any known presence or history of hypogeusia, abnormal taste or dysgeusia;
3. Any known presence or history of severe allergies, or known to be allergic to the components of the test drug;
4. Use of any drugs, including prescription drugs, over-the-counter drugs or herbal preparations, cannot be avoided or expected to start 2 weeks (or 5 half-lives) before screening and throughout the study period;
5. Any findings of electrocardiogram outside from normal, such as the QT interval (QTcF) corrected by the Fridericia formula, the absolute value of QTcF for males is >450 ms, and the absolute value of QTcF for females is >470 ms;
6. Any findings of blood pressure or pulse in resting state outside from normal a: such as systolic blood pressure <90 mmHg or ≥140 mmHg, diastolic blood pressure <60 mmHg or ≥90 mmHg, pulse <55 bpm or >100 bpm;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Number and severity of treatment emergent adverse events | up to 15 days
  Safety and Tolerability Evaluation
Number of participants experiencing AE with abnormal laboratory values | up to 15 days
  Safety and Tolerability Evaluation
Number of participants experiencing AE with abnormal Electrocardiograph | up to 15 days
  Safety and Tolerability Evaluation
Safety and Tolerability Evaluation | up to 15 days
  Number of participants experiencing AE with abnormal vital sign

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | up to 192 hours after the last dose
  To assess Cmax of Multiple ascending oral doses of HS-10383
Area under the curve (AUC) | up to 192 hours after the last dose
  o assess AUC of Multiple ascending oral doses of HS-10383
Time of Maximum Concentration (Tmax) | up to 192 hours after the last dose
  To assess Tmax of Multiple ascending oral doses of HS-10383

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong provincial qianfoshan hospital, Jinan, Shandong, China